CLINICAL TRIAL: NCT02518204
Title: Validity of an Online Neurocognitive Test Battery, the Brain Performance Test (BPT), in Normal Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lumos Labs, Inc. (Industry)
Collaborators: Collaborative Neuroscience Network (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: LL001
Record Dates: First submitted 2015-08-04; First posted 2015-08-07 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Healthy Volunteers
Keywords: cognitive assessment; neuropsychological assessment; Brain Performance Test; computerized assessment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- BPT, NP (Experimental): Computerized assessment battery, followed by a 10 minute break, followed by conventional in-person neuropsychological assessments
  Interventions: Other: BPT; Other: NP
- NP, BPT (Experimental): Conventional in-person neuropsychological assessments, followed by a 10 minute break, followed by a computerized assessment battery
  Interventions: Other: BPT; Other: NP

INTERVENTIONS:
Other: BPT — Brain Performance Test (BPT) computerized cognitive assessment battery developed by Lumos Labs, Inc.
Other: NP — Conventional in-person Neuropsychological Assessments (NP)
  Subtests from:
  * HRB: Halstead-Reitan Battery
  * MATRICS: Measurement and Treatment Research to Improve Cognition in Schizophrenia
  * WAIS-IV: Weschler Adult Intelligence Scale - IV

SUMMARY:
The purpose of this study is to evaluate the concurrent validity between the Brain Performance Test (BPT) subtests and corresponding conventional in-person neuropsychological assessments (NP).

DETAILED DESCRIPTION:
This will be a multi-site, randomized, counterbalanced, two-period, two-sequence, validation study of the online, unsupervised Brain Performance Test (BPT). Over the course of 14 days, participants will complete two in-clinic visits during which they will complete both the BPT and in-person neuropsychological assessments (NP).

ELIGIBILITY:
Inclusion Criteria:

* Native English speaker
* Capable and willing to provide informed consent
* Able to use a computer and mouse without assistance
* Limited (< 3 days) or no experience with Lumosity.com
* Limited (< 3 days) or no experience with other cognitive training programs (e.g., FitBrains, CogMed)
* Willing to refrain from online cognitive training during the course of the study
* No recent (<1 years) experience with either computer-based or in-person neuropsychological tests (e.g., WAIS-IV, WISC, Halstead-Reitan Battery, MATRICS, CogState, CNS Vital Signs)
* Good general health assessed via self-reported online physical questionnaire and medical history questionnaire

Exclusion Criteria:

* Illiterate or unable to understand written English sufficiently to comprehend study instructions and consent form
* Uncorrected visual impairment (beyond that required to qualify for a California Driver's License) that may impact the ability to complete assessments (self-report or determined by the clinician)
* Uncorrected auditory impairment that may impact the ability to complete assessments (self-report or determined by the clinician)
* Self-reported clinical diagnosis for primary psychiatric or neurological disorder (e.g., schizophrenia, multiple sclerosis, attention deficit hyperactivity disorder, Parkinson's disease, epilepsy)
* Self-reported history of concussion or traumatic brain injury, that is considered clinically significant in the opinion of the investigator (e.g. loss of consciousness ≤ 30 minutes)
* Self-reported diagnosis of mental retardation or pervasive developmental disorder
* Self-reported diagnosis of Mild Cognitive Impairment, Alzheimer's disease, or other dementia
* Self-reported history of sustained substance or alcohol abuse or dependence, that is considered clinically significant in the opinion of the investigator (e.g. as defined by DSM-5)
* Self-report that subject is currently taking an antipsychotic, antidepressant, anti-anxiety, or a cognitively-enhancing medication (e.g. Ritalin), or in the last 72 hours, narcotics for pain or other medications that may impact cognitive performance (e.g. sleeping medications/aides or cold/allergy medications)
* Any other significant medical condition that could impact cognitive performance or result in cognitive impairment in the opinion of the investigator
* Score <28 on the MMSE
* Positive urine test for recent substance use on either testing day
* Breath Alcohol Content of 0.01% or greater on either testing day

Ages: 70 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 229 (Actual)
Dates: Start 2015-07; Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Correlation coefficients (Pearson's r) of scaled scores of BPT subtests compared to scaled scores of their NP correlates at Time 1 | 1 day

SECONDARY OUTCOMES:
Interclass correlations (ICC) of scaled scores of BPT subtests compared to scaled scores of their NP correlates at Time 1 | 1 day
Correlation coefficients (Pearson's r and ICC) of raw scores of BPT subtests compared to raw scores of their NP correlates at Time 1 | 1 day
Correlation coefficients (Pearson's r and ICC) of BPT composite indices and NP composite indices at Time 1 | 1 day
Correlation coefficients (Pearson's r and ICC) of raw and scaled scores of BPT subtests at Time 1 and Time 2 as measures of test-retest reliability | 2 weeks
Correlation coefficients (Pearson's r and ICC) of composite indices of BPT and NP at Time 1 and Time 2 as measures of reliability | 2 weeks
Correlation coefficients (Pearson's r and ICC) of BPT Grand Index and NP Overall Index at Time 1 and Time 2 as measures of reliability | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Walling, PhD, Principal Investigator — Collaborative Neuroscience Network
Locations (3):
- United States (3):
  - Orange County Research Center, Garden Grove, California
  - Northern California Research Center, Oakland, California
  - South Bay Research Center, Torrance, California